CLINICAL TRIAL: NCT03781739
Title: A PHASE I, DOUBLE BLIND, PLACEBO-CONTROLLED STUDY EVALUATING THE CARDIOVASCULAR AND METABOLIC PROPERTIES OF MANP IN SUBJECTS WITH HYPERTENSION AND METABOLIC SYNDROME ACCORDING TO RS5068 GENOTYPES
Brief Title: MANP in Hypertension and Metabolic Syndrome
Acronym: MANP-HTN-MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Paul M. McKie, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB # 16-005813
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Hypertension; Metabolic Syndrome
MeSH Terms: conditions — Hypertension; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MANP (Experimental): subjects receiving MANP (2.5 micrograms/kg, single subcutaneous injection)
  Interventions: Drug: MANP
- Placebo (Placebo Comparator): subjects receiving placebo (saline solution, single subcutaneous injection)
  Interventions: Drug: MANP

INTERVENTIONS:
Drug: MANP — single subcutaneous injection of MANP and monitoring of metabolic, cardiovascular and renal parameters

SUMMARY:
Evaluate the cardiovascular and metabolic properties of MANP in subjects with HTN and MS according to rs5068 genotypes

DETAILED DESCRIPTION:
6 Study Procedures 6.1 Day 0 - Visit 1 (screening visit) 6.2 At visit 1 informed consent will be obtained (Table 1). Introduction and orientation to the study will take place. Medical history will be collected. Physical exam will be performed and laboratory exams history will be screened. Electrocardiogram will be recorded and screening laboratory tests will be performed. Blood pressure and heart rate will be recorded. Subjects will be instructed about the fluid intake allowed (2.5 liter/day) and the diet (moderate sodium intake: 3.0 gr/day) to follow for the duration of the study from day 1 to day 7. Subjects will be instructed on completing a 24-hour urine collection starting on day 4 at 4pm (see day 4 below). Antihypertensive medications are required to be at a stable dose for 30 days preceding visit 1 on day 1. Throughout the duration of the study subjects will be maintained on their chronic antihypertensive treatment except for day 6 in which MANP or placebo will be administered. Subjects will be instructed to avoid strenuous physical activities and to abstain from smoking and alcohol from day 1 until the completion of the study on day 7. Caffeine consumption will be prohibited from 7.00 pm on day 5 until the dismissal from the CRTU on day 7. Day 1 Start of diet and fluid restriction compliance. (Interval of time between day 0 and day 1 will depend upon the CRTU schedules 6.3 Day 4 On Day 4 at 4 pm the subjects will start 24-hour urine collection in order to establish adherence to the moderate sodium diet (Table 1).

6.4 Day 5 On day 5 at 4pm subjects will bring the 24-hour urine collection to the CRTU and 24-hour urine sodium will be measured. If the patient has been compliant with the sodium diet, she/he will be admitted to the CRTU to continue the study and a physical exam will be performed. At 7.00 pm subjects will start fasting and abstain from their usual hypoglycemic therapy in consideration of the blood draws for metabolic parameters that will be performed on day 6. Caffeine consumption is prohibited from 7:00 pm on day 5 until the dismissal from the CRTU on day 7.

6.5 Day 6 - Visit 2 On day 6 at 8:00 am enrolled patients will receive a single injection of MANP (2.5 μg/kg SQ) or placebo (0.9% saline solution) and will be under observation for the 24 hours following the MANP/placebo administration (Table 1). Blood pressure and heart rate will be monitored continually and recorded before MANP/placebo injection and at several intervals after MANP/placebo administration. Timed urine collection and blood samples to evaluate neurohumoral, renal function and metabolic plasma parameters will be collected prior to MANP /placebo injection and at different time points after MANP and placebo administration. Subjects will eat their meal and take their usual hypoglycemic medications after the last blood draw for metabolic parameters (4 hours after the MANP injection). Subjects will be maintained on their chronic antihypertensive treatment except for day 6 in which MANP will be administered. They will take their usual antihypertensive therapy 24 hours after MANP injection.

6.6 Day 7 Once completed the 24 hour observation following MANP administration a physical exam will be performed and the subjects will be dismissed from the CRTU

6.7 Day 14 (± 2 days) Laboratory tests will be performed and assessed. Subjects will be contacted by phone to review laboratory tests results and assess the onset of any potential side effect following the MANP/placebo administration.

6.8 Day 30 (-2 days, + 5 days) Blood collection for anti-MANP antibody testing will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension defined as 140 mmHg ≤ systolic BP ≤ 180 mmHg or 90 mmHg ≤ diastolic BP ≤ 100 mmHg despite anti-hypertensive medical therapy
* Metabolic Syndrome defined as the presence of any two of the following traits:
* Abdominal obesity, defined as a waist circumference in men ≥102 cm (40 in) and in women ≥88 cm (35 in)
* Serum triglycerides ≥150 mg/dL (1.7 mmol/L)
* Serum HDL cholesterol <40 mg/dL (1 mmol/L) in men and <50 mg/dL (1.3 mmol/L) in women or drug treatment for low HDL cholesterol
* Fasting plasma glucose ≥100 mg/dL (5.6 mmol/L) or drug treatment for elevated blood glucose
* Between the ages of 18 and 75 years
* Use of antihypertensive medications at a stable dose for 30 days preceding screening visit.
* Use of statins or ezetimibe or combinations on stable dose for 60 days preceding screening visit.

Exclusion Criteria:

* Known hypersensitivity or allergy to MANP or its components, carperitide, other natriuretic peptides, or related compounds;
* Subjects with orthostatic hypotension at the screening visit, defined as a decrease in systolic BP of >20 mmHg or a decrease in diastolic BP of >10 mmHg within three minutes of standing when compared with blood pressure from the sitting position.
* Subjects with a systolic BP >180 mmHg or a diastolic BP >100 mmHg
* Women of child-bearing potential
* The presence of abnormal laboratory values at screening visit considered clinically significant by the Investigator. Specifically they will be excluded if a) Serum sodium of < 135 mEq/dL or > 145 mEq/dL; b) Serum potassium of < 3.5 mEq/dL or > 5.1 mEq/dL
* Subjects whose body weight has changed more than 3% in the last 3 months
* Having received any investigational drug or device within 30 days prior to entry into the study;
* A history (within the last 2 years) of alcohol risky use (defined as more than 14 standard drinks per week on average or more than 4 drinks on any day for men under age 65 - defined as more than 7 standard drinks per week on average or more than 3 drinks on any day for women and adults 65 years and older);
* A history of illicit drug use, psychiatric illness that might impair the participation to the study, physical dependence to any opioid, or any history of substance abuse or addiction;
* A history of difficulty with donating blood or donated blood or blood products within 45 days prior to enrollment;
* Clinically significant new illness in the 1 month before screening in the opinion of the Investigator;
* History of severe allergies;
* History of coronary artery disease or cerebrovascular disease or syncope;
* History of epilepsy or other seizure disorder;
* History of organ transplantation;
* Malignancy within 5 years of the screening visit (with the exception of basal cell and squamous cell skin carcinoma);
* Clinically significant intrinsic renal disease, renal artery stenosis, or history of fibromuscular dysplasia of the renal arteries;
* Consumption of a phosphodiesterase-5 inhibitor (sildenafil, vardenafil, or tadalafil) within 72 hours of receiving MANP.
* Episodic or chronic use of nitrates (Isordil, nitroglycerine), MAO inhibitors, antipsychotics, antiarrhythmics, psychostimulants, systemic corticosteroids, cholestyramine and cholestipol reisins, fibrates, nicotinic acid, cyclosporin, rifampin or other highly potent PgP inhibitors.
* Any disease or condition (medical or surgical) which, in the opinion of the investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk.
* Subjects who smoke or have any history of tobacco product use more recently than 6 months prior to the enrollment into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
cardiovascular outcome | 24 hours
  systolic blood pressure
second messenger | 24 hours
  cGMP plasma levels
metabolic outcome | 24 hours
  glycerol and non-esterified fatty acids (NEFA) plasma levels

SECONDARY OUTCOMES:
secondary cardiovascular outcome | 24 hours
  diastolic blood pressure
secondary metabolic outcome | 24 hours
  adiponectin plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Paul M McKie, M.D., Principal Investigator — Mayo Foundation
Locations (1):
- Mayo Foundation, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma X, McKie PM, Iyer SR, Scott C, Bailey K, Johnson BK, Benike SL, Chen H, Miller WL, Cabassi A, Burnett JC Jr, Cannone V. MANP in Hypertension With Metabolic Syndrome: Proof-of-Concept Study of Natriuretic Peptide-Based Therapy for Cardiometabolic Disease. JACC Basic Transl Sci. 2023 Nov 1;9(1):18-29. doi: 10.1016/j.jacbts.2023.08.011. eCollection 2024 Jan. PMID 38362338
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials